CLINICAL TRIAL: NCT03422952
Title: Hormonal and Physiological Stress Response of Medical Doctors Working in Rescue Helicopter or Van
Brief Title: Stress Response in Emergency Among Physicians in Helicopter and Ambulance Based Emergency Medical Systems
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00561
Record Dates: First submitted 2017-05-15; First posted 2018-02-06 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Hormone Disturbance; Stress Reaction; Stress Related Disorder
MeSH Terms: conditions — Endocrine System Diseases; Fractures, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Cortisol
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stress reactions in emergency physicians will be measures using cortol-awakening-reaction, heart-rate-variability and standardised stress questionnaires

DETAILED DESCRIPTION:
In a field study with within-subject design, there will be conducted the hormonal and physiological stress strain of emergency physicians working in rescue helicopters or van on different days of service on different headquarters. The investigation of the parameter of stress will be conducted on two days of rescue service, on two days of clinical service and as a control on two days off. The quantification of the hormonal stress strain will be carried out with the cortisol awakening response, there will be conducted 3 saliva samples with identical interval after getting up within 30 minutes. While the labour time on the rescue service and on the clinical service and the whole day off, the heart rate variability will show the degree of physiological stress. This will be measured with a pulse-belt on the chest, which the participant will carry the whole day. In addition, participants will fill out a set of questionnaire on the first day of measurement.

ELIGIBILITY:
Inclusion Criteria:

* Medical Doctor working in rescue helicopter or van

Exclusion Criteria:

* Metabolic disease
* Autoimmune disease
* Heart disease
* Blood disease
* Mental disease
* Endocrinologic disease
* BMI>30
* >10 cigarettes/day
* Taking cortisone medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical Doctor working in rescue helicopter or van
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Cortisol-awakening-response (CAR) | 30 min each day, six days
  Differences on the CAR on rescue services, clinical services and on days off.
Heart rate variability | six days
  Continuous measurement
Stress questionnaire | first day
  Subjective perceived strain with questionnaires with validated scores of stress

OTHER OUTCOMES:
Possible factors that may affect the measured parameter | six days
  Monitoring the health status and workload:
  BMI kg/m2 Heartrate bpm Bloodpressure mmHg Body-Temperature °C Time working h

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Theiler, PD Dr. med, Principal Investigator — attending anaesthesiologist
Locations (1):
- Bern University Hospital and University of Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No